CLINICAL TRIAL: NCT02502812
Title: An Open-label, Randomised, Single-dose, Three-way Cross Over, Six Sequence Study to Determine the Relative Bioavailability of Clopidogrel 75mg From Two Tablet Formulations of SB224326 Relative to One 75mg Reference Tablet of Clopidogrel in Healthy Adult Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Clopidogrel 75 mg in Two Tablet Formulations Relative to Reference Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200096
Record Dates: First submitted 2015-07-09; First posted 2015-07-20 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Cardiovascular Disease
Keywords: bioequivalence; SB224326; clopidogrel; Relative bioavailability
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment Sequence A (Innovator) - B (Clop F1) - C (Clop F2) (Experimental): Subjects will receive a single 75 mg tablet of reference clopidogrel (Treatment A) in treatment period 1, 75 mg tablet Clop F1 (Treatment B) in treatment period 2, and 75 mg tablet Clop F2 (Treatment C) in treatment period 3 under fasting conditions. Each treatment period will be separated by 7-14 days of washout Period.
  Interventions: Drug: Clop F1; Drug: Clop F2; Drug: Innovator
- Treatment Sequence A(Innovator) -C(Clop F2)-B (Clop F1) (Experimental): Subjects will receive a single 75 mg tablet of reference clopidogrel (Treatment A) in treatment period 1, 75 mg tablet Clop F2 (Treatment C) in treatment period 2, and 75 mg tablet Clop F1 (Treatment B) in treatment period 3 under fasting conditions. Each treatment period will be separated by 7-14 days of washout Period.
  Interventions: Drug: Clop F1; Drug: Clop F2; Drug: Innovator
- Treatment Sequence B (Clop F1) - A (Innovator) - C (Clop F2) (Experimental): Subjects will receive a single 75 mg tablet Clop F1 (Treatment B) in treatment period 1, 75 mg tablet of reference clopidogrel (Treatment A) in treatment period 2, and 75 mg tablet Clop F2 (Treatment C) in treatment period 3 under fasting conditions. Each treatment period will be separated by 7-14 days of washout Period.
  Interventions: Drug: Clop F1; Drug: Clop F2; Drug: Innovator
- Treatment Sequence B (Clop F1) - C (Clop F2) - A (Innovator) (Experimental): Subjects will receive a single 75 mg tablet Clop F1 (Treatment B) in treatment period 1, 75 mg tablet Clop F2 (Treatment C) in treatment period 2, and 75 mg tablet of reference clopidogrel (Treatment A) in treatment period 3 under fasting conditions. Each treatment period will be separated by 7-14 days of washout Period.
  Interventions: Drug: Clop F1; Drug: Clop F2; Drug: Innovator
- Treatment Sequence C (Clop F2) - A (Innovator) - B (Clop F1) (Experimental): Subjects will receive a single 75 mg tablet Clop F2 (Treatment C) in treatment period 1, 75 mg tablet of reference clopidogrel (Treatment A) in treatment period 2, and 75 mg tablet Clop F1 (Treatment B) in treatment period 3 under fasting conditions. Each treatment period will be separated by 7-14 days of washout Period.
  Interventions: Drug: Clop F1; Drug: Clop F2; Drug: Innovator
- Treatment Sequence C (Clop F2) - B (Clop F1) - A (Innovator) (Experimental): Subjects will receive a single 75 mg tablet Clop F2 (Treatment C) in treatment period 1, 75 mg tablet Clop F1 (Treatment B) in treatment period 2, and 75 mg tablet of reference clopidogrel (Treatment A) in treatment period 3 under fasting conditions. Each treatment period will be separated by 7-14 days of washout Period.
  Interventions: Drug: Clop F1; Drug: Clop F2; Drug: Innovator

INTERVENTIONS:
Drug: Clop F1 — A single oral dose of clopidogrel (bisulfate) 75 mg tablet will be administered with approximately 240 mL water in fasted state.
Drug: Clop F2 — A single oral dose of clopidogrel (bisulfate) 75 mg tablet will be administered with approximately 240 mL water in fasted state.
Drug: Innovator — A single oral dose of clopidogrel (bisulfate) 75 mg tablet will be administered with approximately 240 mL water in fasted state.

SUMMARY:
Clopidogrel is a potent anti-thrombotic drug that inhibits adenosine diphosphate (ADP)-induced platelet aggregation. This is an open-label, randomized, single dose, three-way cross over, six sequence study to investigate the relative bioavailability of two 75 milligrams (mg) clopidogrel tablet formulations (clopidogrel SB224326 test formulation 1 [Clop F1] and clopidogrel SB224326 test formulation 2 [Clop F2]) compared with the reference product (innovator) in healthy human subjects. A total of 18 healthy human subjects will be randomized, such that approximately 14 evaluable subjects complete the study. Total duration in the study for each subject will be approximately 8 weeks from screening to the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy, non-smoker, as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilograms (kg) and Body mass index (BMI) within the range 19 - 24.9 kg/square meter (m^2) (inclusive).
* Healthy male or female subjects: MALES: Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until 24 hours after the last dose of study medication: a) Vasectomy with documentation of azoospermia. b) Male condom plus partner use of one of the contraceptive following options: Contraceptive subdermal implant, Intrauterine device or intrauterine system, Oral Contraceptive, either combined or progestogen alone, Injectable progestogen, Contraceptive vaginal ring, Percutaneous contraceptive patches, This is an all inclusive list of those methods that meet the GlaxoSmithKline (GSK) definition of highly effective: having a failure rate of less than 1% per year when used consistently and, correctly and, when applicable, in accordance with the product label. For non-product methods (e.g. male sterility), the investigator determines what is consistent and correct use. The GSK definition is based on the definition provided by International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH). The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception. FEMALES: Eligible to participate, if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies: a) Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy, Postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. b) Reproductive potential and agrees to follow one of the options listed below in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until 24 hours after the last dose of study medication and completion of the follow-up visit.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Innovator product contains lactose and subjects with lactose intolerance should not be included.
* Alanine aminotransferase (ALT) and bilirubin >1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Corrected QT interval (QTc) > 450 milliseconds (msec) NOTES: The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read. The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial. For purposes of data analysis, QTcB, QTcF, another QT correction formula, or a composite of available values of QTc will be used.
* The following medications increase risk of bleeding: Nonsteroidal anti-inflammatory drugs (NSAIDs), warfarin, selective serotonin and serotonin norepinephrine reuptake inhibitors (SSRIs, SNRIs).
* Proton pump inhibitors: some drugs from this class have an inhibitory effect on the formation of clopidogrel active metabolite.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (~240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Active pathological bleeding, such as peptic ulcer or intra cranial haemorrhage
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Gastrointestinal disease or with gastrointestinal surgical history which can affect the absorption of the investigational drug.
* Any symptoms with a systolic blood pressure (BP) <95 millimeter of mercury (mmHg)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09-04 (Actual); Primary Completion 2015-09-24 (Actual); Study Completion 2015-09-24 (Actual)

PRIMARY OUTCOMES:
Composite of plasma pharmacokinetic (PK) parameters: AUC(0 ∞), AUC(0 t) and Cmax | Day 1: pre-dose, 0.25, 0.5, 0.75, 1.00, 1.33, 1.67, 2, 2.5, 3.00, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00 (Day 2) hours post-dose of each treatment period
  The following PK parameters were measured: area under the plasma concentration-time curve from time zero to infinity (AUC[0 ∞]), area under the plasma concentration-time curve from time zero to last time point with measurable concentration (AUC[0 t]) and maximum observed plasma concentration (Cmax)

SECONDARY OUTCOMES:
Composite of plasma PK parameters: time of occurrence of Cmax (tmax), percentage of AUC(0 ∞) obtained by extrapolation (%AUCex) and terminal phase half-life (t1/2) | Day 1: pre-dose, 0.25, 0.5, 0.75, 1.00, 1.33, 1.67, 2, 2.5, 3.00, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00, 24.00 (Day 2) hours post-dose of each treatment period
  Pre-dose PK blood samples will be collected within 60 minutes prior to dose. Post dose blood samples will be collected within 2 minutes.
Blood pressure as a measure of safety and tolerability | Up to 8 weeks
  Blood pressure will be measured at predose, 0.50, 1.00, 2.00, 4.00, and 24.00 hours post-dose. Post dose blood pressure to be taken plus or minus 30 minutes of each timepoint.
Pulse rate as a measure of safety and tolerability | Up to 8 weeks
  Pulse rate will be measured at predose, 0.50, 1.00, 2.00, 4.00, and 24.00 hours post-dose. Post dose pulse rate to be taken plus or minus 30 minutes of each timepoint.
Number of subjects with adverse events and serious adverse events | From start of study medication until follow up (Up to 5 weeks)
  An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE was defined as any untoward medical occurrence that, at any dose, resulted in death, was life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect, or was an event of possible drug-induced liver injury.
Composite of hematology parameters as a measure of safety | Up to 8 weeks
  The following hematology assessments will be performed: platelet count, red blood cell (RBC) count, hemoglobin, hematocrit, white blood cells (WBC) (absolute), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), neutrophils, lymphocytes, monocytes, eosinophils, and basophils.
Composite of clinical chemistry parameters as a measure of safety | Up to 8 weeks
  The following clinical chemistry assessments will be performed: blood urea nitrogen (BUN), creatinine, fasting glucose, potassium, sodium, calcium, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, total and direct bilirubin, total protein, and albumin.
Composite of urinalysis parameters as measured by dipstick method and microscopic examination | Up to 8 weeks
  Dipstick method will be used to measure pH, glucose, protein, blood and ketones. Microscopic examination will be performed if blood or protein is abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Telangana, India

REFERENCES:
- See also: Results for study 200096 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/200096?search=study&b'search_terms=200096'#rs